CLINICAL TRIAL: NCT06750068
Title: Clinical Evaluation of Digitally Fabricated 3D-printed Band and Loop Space Maintainers Versus Conventional Band and Loop Space Maintainer : a Randomized Clinical Trial
Brief Title: Evaluation of 3D-printed Space Maintainers Versus Conventional Space Maintainer : a Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Alaa Abdelaziz Elsayed, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 16111992ayaalaaabdelazizelsaye
Record Dates: First submitted 2024-12-16; First posted 2024-12-27 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-12

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Intervention Model Description: 3D printed band and loop space maintainer Conventions band and loop space maintainer
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional band and loop space maintainer (Active Comparator): Impressions will be taken from the patients with sterilized plastic pedodontic impression trays and alginate under standard conditions by the same researcher. Alginate will be mixed in accordance with the manufacturer's instructions. After the impressions, plaster study casts will be produced and sent to the laboratory. Conventional SMs will be produced by soldering the 0.7-mm bent orthodonic wires (Dentaurum, Germany) onto previously selected prefabricated molar bands. Prefabricated molar bands (Dentaurum, Germany) in the patient's mouth will be chosen by the physician and then sent to the laboratory with the casts.
  All SMs will be cemented by the same investigator under standard conditions using a glass-ionomer luting cement (Nova Glass-L, Imicryl, Konya, Turkey).
  Interventions: Other: Conventional space maintainer
- 3D printed space maintainer (Experimental): Patients in this group will be scanned under standard conditions with Medit i500 (Medit Corp. Seoul, South Korea). The scanned data of the patients will be sent to the laboratory via email in Standard Triangle Language (STL) file format.The design of SMs will be carried out on the DentalCAD 2.2 Valletta (Exocad GmbH, Darmstadt, Germany) program to mimic the conventional space maintainer, and the production will be made by the 3D Selective laser melting (SLM Solutions, Germany) method using titanium-based metal powder (Ti64 Gd23; LPW Technology Ltd., Cheshire, UK). The production of 3D-SMs will start in accordance with the C-SM design in many points, such as the fit of the part surrounding the abutment tooth, thickness, and the position of the loop of 3D-SM.
  All SMs will be cemented by the same investigator under standard conditions using a glass-ionomer luting cement (Nova Glass-L, Imicryl, Konya, Turkey).
  Interventions: Other: 3D printed space maintainer

INTERVENTIONS:
Other: 3D printed space maintainer — Digitally fabricated #d printed space maintainer
  Arms: 3D printed space maintainer
Other: Conventional space maintainer — Stainless steel space maintains
  Arms: Conventional band and loop space maintainer

SUMMARY:
This study aims to compare the clinical evaluation and patients' satisfaction of space maintainers produced by digital workflow using the 3D-printing method (3D-SMs) versus conventional band and loop space maintainers (C-SMs) produced by traditional methods.

ELIGIBILITY:
Inclusion Criteria:

* Lower first permanent molar in active state of eruption
* Patient and parent showing cooperation and compliance.
* Medically free children.
* According to space analysis available space is less than or equal to needed space
* Primary molar loss in the last 1 week due to caries, infection, and resorption (to eliminate possible space loss)
* Caries free, non-restored buccal surfaces of the mandibular second primary molars and deciduous canines.

Exclusion Criteria:

* Children with previous allergies to stainless steel.
* There was less than one year left for the permanent tooth to erupt (to prevent possible abutment toot loss)
* The patient's oral hygiene is not sufficient and has periodontal problems (to accurately assess the periodontal effects)

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 1 year
  Decementation, debonding, solder breakage, loop breakage, band breakage, and abutment tooth fracture will be evaluated clinically for both space maintainers

SECONDARY OUTCOMES:
Gingival health of the abutment | 0,6,12 months
  Gingival index 0 = normal gingiva; 1 = mild inflammation: slight change in color, slight edema, no bleeding on probing; 2 = moderate inflammation: redness, edema, and glazing, or bleeding on probing; 3 = severe inflammation: marked redness and edema, tendency toward spontaneous bleeding
Plaque accumulation on the abutment tooth | 0,6,12 months
  Plaque index Score 0: No Plaque Score 1:Thin plaque layer at the gingival margin, only detectable by scraping with a probe Score 2: Moderate layer of plaque along the gingival margin; interdental spaces free, but plaque is visible to the naked eye Score 3:Abundant plaque along the gingival margin; interdental spaces filled with plaque
Patients' satisfaction about the impression technique | Immediately after the im- pression/scanning
  Five- question survey
  1. "Was the impression easy and fun?"
  2. "Did you have nausea during impression?"
  3. "Did you feel any discomfort during the impression (taste, odor, foreign body)?"
  4. "Did the impression take a short time?"
  5. "Would you like to have this impression experience again?"

IPD SHARING:
Plan to Share IPD: No